CLINICAL TRIAL: NCT05349617
Title: A Phase 3 Safety and Immunogenicity Trial of the VLP-Based Chikungunya Virus Vaccine PXVX0317 in Adults ≥65 Years of Age
Brief Title: Safety and Immunogenicity of CHIKV VLP Vaccine PXVX0317 in Adults ≥65 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Collaborators: Emergent BioSolutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EBSI-CV-317-005
Record Dates: First submitted 2022-04-21; First posted 2022-04-27 (Actual); Results first posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Chikungunya Virus
Keywords: chikungunya; virus like particle (VLP); PXVX0317; vaccine; immunogenicity
MeSH Terms: conditions — Chikungunya Fever

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio to receive PXVX0317 or placebo within each age stratum. Participants will be stratified in two age subgroups (≥65 to <75 and ≥75 years of age). This study will be conducted in the US, using up to 10 sites.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 - PXVX0317 (Experimental): PXVX0317 vaccine is comprised of chikungunya virus virus-like particles (CHIKV VLP), adsorbed on aluminum hydroxide adjuvant.
  Interventions: Biological: CHIKV VLP/adjuvant
- Group 2 - Placebo (Placebo Comparator): Placebo is comprised of formulation buffer.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CHIKV VLP/adjuvant — PXVX0317 vaccine is comprised of chikungunya virus virus-like particles (CHIKV VLP), adsorbed on aluminum hydroxide adjuvant
  Arms: Group 1 - PXVX0317
Biological: Placebo — Placebo is comprised of formulation buffer
  Arms: Group 2 - Placebo

SUMMARY:
The purpose of this phase 3, randomized, double-blind, placebo-controlled study is to evaluate the safety and immunogenicity to PXVX0317 in adults ≥65 years of age.

DETAILED DESCRIPTION:
Co-primary Objectives:

* To compare the anti-CHIKV serum neutralizing antibody (SNA) response to PXVX0317 and placebo at Day 22, as measured by geometric mean titer (GMT) and clinically relevant difference in seroresponse rate (PXVX0317 minus placebo) in adults ≥65 years of age.
* To evaluate the safety of PXVX0317 in adults ≥65 years of age

Secondary Objectives:

* To compare the anti-CHIKV SNA response to PXVX0317 and placebo at Day 15 and Day 183, as measured by GMT and seroresponse rate.
* To compare the anti-CHIKV SNA response to PXVX0317 and placebo in participants ≥65 to <75 and ≥75 years of age as measured by GMT and seroresponse rate.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide informed consent voluntarily signed by participant. Must verbalize understanding of the general procedures of, and reason for the study.
* Males or females, ≥65 years of age.
* Able to complete all scheduled visits and comply with all study procedures.
* Women who are not of childbearing potential (CBP): surgically sterile (at least six weeks post bilateral tubal ligation, bilateral oophorectomy or hysterectomy); or postmenopausal (defined as a history of ≥12 consecutive months without menses prior to randomization in the absence of other pathologic or physiologic causes, following cessation of exogenous post menopausal sex-hormonal treatment).
* Participants must be in stable health in the opinion of the investigator for at least 30 days prior to screening (eg, no hospital admission for acute illness in the last 30 days prior to screening).

Exclusion Criteria:

* Participation or planned participation in an investigational clinical trial (eg, vaccine, drug, medical device, or medical procedure) within 30 days of Day 1 and for the duration of the study. Note: Participation in an observational trial or follow-up phase of a trial may be allowed; however, these instances should be discussed with the sponsor's medical monitor (MM) prior to enrollment.
* Prior receipt of any CHIKV vaccine.
* Positive laboratory evidence of current infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV) or hepatitis B virus (HBV).
* Body mass index (BMI) ≥35 kg/m^2
* History of any known or suspected allergy or history of anaphylaxis to any component of the investigational product (IP).
* History of any known congenital or acquired immunodeficiency or immunosuppressive condition that could impact response to vaccination (eg, leukemia, lymphoma, malignancy, functional or anatomic asplenia, alcoholic cirrhosis). Note: History of basal cell and squamous cell carcinoma of the skin or carcinoma in situ of the cervix considered cured would not be exclusionary. History of a malignancy considered cured from over five years from the date of screening with minimal risk of recurrence is not exclusionary.
* Prior or anticipated use of systemic immunomodulatory or immunosuppressive medications from six months prior to screening through Day 22. Note: Systemic corticosteroid use at a dose or equivalent dose of 20 mg of prednisone daily for 14 days or more within 90 days of screening through Day 22 is exclusionary. The use of inhaled, intranasal, topical, or ocular steroids is allowed.
* Bleeding disorder or receipt of anticoagulants in the 21 days prior to screening, contraindicating intramuscular (IM) vaccination, as judged by the investigator.
* Moderate or severe acute illness with or without fever (oral temperature ≥100.4°F or 38.0°C).
* Receipt or anticipated receipt of immunoglobulin from 180 days prior to screening through Day 22.
* Medical condition (such as dementia) that, in the opinion of the investigator, could adversely impact the participant's participation in or conduct of the study.
* Evidence of substance abuse that, in the opinion of the investigator, could adversely impact the participant's participation in or conduct of the study.
* Identified as an investigator or employee of an Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (ie, parent, spouse) of the investigator or employee with direct involvement in the proposed study.
* Receipt or anticipated receipt of any vaccine from 30 days prior to Day 1 through Day 22.
* Receipt or anticipated receipt of blood or blood-derived products from 90 days prior to screening through Day 22.
* Any planned elective surgery that may interfere with study participation or conduct.
* Any other medical condition that, in the opinion of the investigator, could adversely impact the participant's participation in or conduct of the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 413 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Ajiboye, MD, Study Director — Bavarian Nordic
Locations (10):
- United States (10):
  - Suncoast Research Associates, LLC, Miami, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - Global Clinical Research Professionals (GCP), St. Petersburg, Florida
  - AMR Kansas City, Kansas City, Missouri
  - Rochester Clinical Research, Inc., Rochester, New York
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - DM Clinical Research CyFair, Houston, Texas
  - BHFC Research, San Antonio, Texas
  - DM Clinical Research Tomball, Tomball, Texas
  - Spaulding Clinical, West Bend, Wisconsin

REFERENCES:
- [Derived] Tindale LC, Richardson JS, Anderson DM, Mendy J, Muhammad S, Loreth T, Tredo SR, Ramanathan R, Jenkins VA, Bedell L, Ajiboye P; EBSI-CV-317-005 Study Group. Chikungunya virus virus-like particle vaccine safety and immunogenicity in adults older than 65 years: a phase 3, randomised, double-blind, placebo-controlled trial. Lancet. 2025 Apr 19;405(10487):1353-1361. doi: 10.1016/S0140-6736(25)00372-1. Epub 2025 Mar 27. PMID 40158524
- [Derived] Bennett SR, McCarty JM, Ramanathan R, Mendy J, Richardson JS, Smith J, Alexander J, Ledgerwood JE, de Lame PA, Royalty Tredo S, Warfield KL, Bedell L. Safety and immunogenicity of PXVX0317, an aluminium hydroxide-adjuvanted chikungunya virus-like particle vaccine: a randomised, double-blind, parallel-group, phase 2 trial. Lancet Infect Dis. 2022 Sep;22(9):1343-1355. doi: 10.1016/S1473-3099(22)00226-2. Epub 2022 Jun 13. PMID 35709798

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter study conducted in the United States, using 10 sites. Healthy adult participants ≥65 year of age were enrolled in this study. Recruitment Period was from May 12, 2022 to December 02, 2022.
Period: Overall Study
Arm/Group | Group 1 - PXVX0317 | Group 2 - Placebo
Started | 206 | 207
Completed | 200 | 188
Not Completed | 6 | 19
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 3 | 8
Not completed — Withdrawal by Subject | 2 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - PXVX0317 | Group 2 - Placebo | Total
Number analyzed (Participants) | 206 | 207 | 413
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (5.3) | 71 (4.5) | 71 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 117 | 242
  Male | 81 | 90 | 171
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 93 | 90 | 183
  Not Hispanic or Latino | 112 | 116 | 228
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 29 | 49
  White | 176 | 168 | 344
  More than one race | 4 | 5 | 9
  Unknown or Not Reported | 1 | 3 | 4
Height [Mean (Standard Deviation); unit: cm] | 166.4 (9.42) | 167.1 (9.84) | 166.8 (9.63)
Weight [Mean (Standard Deviation); unit: kg] | 75.8 (13.61) | 77.2 (13.29) | 76.5 (13.45)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.3 (3.98) | 27.6 (3.9) | 27.5 (3.94)
Baseline Anti-CHIKV SNA Serostatus [Count of Participants; unit: Participants]
  Negative (<LLOQ) | 201 | 196 | 397
  Positive (≥LLOQ) | 5 | 10 | 15
  Missing | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Anti-CHIKV SNA Titer (NT80) Seroresponse Rates at Day 22 in Baseline Seronegative Participants
Description: Difference in anti-CHIKV SNA titer (NT80) seroresponse rate (PXVX0317 minus placebo) and associated 95 percent confidence interval (CI) at Day 22.
Time Frame: 21 days postvaccination
Population: Immunogenicity Evaluable Population (IEP): All participants in the modified intent-to-treat (mITT) population who provide evaluable serum sample results for Day 22 within the required time frame of Day 19 through Day 27, inclusive; have no measurable anti-CHIKV SNA at Day 1; and have no important protocol deviation or other reason to be excluded as defined prior to unblinding. IEP is the primary population for all immunogenicity analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 - PXVX0317 | Group 2 - Placebo
Number analyzed (Participants) | 189 | 183
percentage of participants | 87.3 [81.8 to 91.3] | 1.1 [0.3 to 3.9]
Statistical Analysis 1: Comparison: Group 1 - PXVX0317 vs Group 2 - Placebo; Day 22; Test type: Superiority; p < 0.0001, Chi-squared — p-value is from a two-sided chi-square test of equality of seroresponse percentages between groups. Both coprimary endpoints were required to be met for success, so no multiple comparisons were performed; Percent Difference = 86.2, 95% CI 2-sided [80 to 90.3] — Seroresponse rate difference is (PXVX0317 minus placebo)

2. Primary Outcome: Anti-CHIKV SNA Titer (NT80) Geometric Mean Titers (GMT) at Day 22
Description: Anti-CHIKV SNA titer (NT80) GMT and associated 95 percent CIs at Day 22 for PXVX0317 and placebo.
Time Frame: 21 days postvaccination
Population: Immunogenicity evaluable population (all randomized and vaccinated participants who provided an evaluable Day 22 anti-CHIKV human SNA assay sample within the analysis window (Day 19 through 27, inclusive), had no measurable anti-CHIKV human SNA assay titer at Day 1 (i.e., seronegative at baseline; participants missing a Day 1 titer were excluded from IEP), and had no important exclusionary protocol deviation or other reason for exclusion as defined prior to unblinding).
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1 - PXVX0317 | Group 2 - Placebo
Number analyzed (Participants) | 189 | 183
Titer | 724 [584 to 897] | 8 [7 to 10]
Statistical Analysis 1: Comparison: Group 1 - PXVX0317 vs Group 2 - Placebo; Day 22; Test type: Superiority; p < 0.0001, ANOVA — Both coprimary endpoints were required to be met for success, so no multiple comparisons were performed; ANOVA model covers site and treatment group as fixed effects, assuming log titers' normality. p-value tests equivalence of mean titers between groups; [GMT Ratio] = 90, 95% CI 2-sided [69 to 117] — Ratio of GMTs is (PXVX0317:placebo)

3. Primary Outcome: Incidence of Solicited Adverse Events (AE)
Description: Incidence of solicited AEs through Day 8 for PXVX0317 (CHIKV VLP vaccine) and placebo for all age strata combined (safety population).
Time Frame: 7 days postvaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - PXVX0317 | Group 2 - Placebo
Number analyzed (Participants) | 205 | 200
Participants | 25 | 28

4. Primary Outcome: Incidence of Unsolicited AEs
Description: Incidence of unsolicited AEs through Day 29 for PXVX0317 (CHIKV VLP vaccine) and placebo for all age strata combined (safety population).
Time Frame: 28 days postvaccination
Population: Safety population (vaccinated participants who provided safety assessment data), All ages pooled.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - PXVX0317 | Group 2 - Placebo
Number analyzed (Participants) | 206 | 207
Participants | 26 | 34

5. Primary Outcome: Incidence of Serious Adverse Events (SAE)
Description: Incidence of SAEs through Day 183 for PXVX0317 (CHIKV VLP vaccine) and placebo for all age strata combined (safety population).
Time Frame: 182 days postvaccination
Population: Safety population (vaccinated participants who provided safety assessment data), All ages pooled.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - PXVX0317 | Group 2 - Placebo
Number analyzed (Participants) | 206 | 207
Participants | 4 | 3

6. Primary Outcome: Incidence of Medically Attended Adverse Events (MAAE)
Description: Incidence of MAAEs through Day 183 for PXVX0317 (CHIKV VLP vaccine) and placebo for all age strata combined (safety population).
Time Frame: 182 days postvaccination
Population: Safety population (vaccinated participants who provided safety assessment data), All ages pooled.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - PXVX0317 | Group 2 - Placebo
Number analyzed (Participants) | 206 | 207
Participants | 19 | 23

7. Primary Outcome: Incidence of Adverse Events of Special Interest (AESI)
Description: Incidence of AESIs, through Day 183 for PXVX0317 (CHIKV VLP vaccine) and placebo for all age strata combined (safety population).
Time Frame: 182 days postvaccination
Population: Safety population (vaccinated participants who provided safety assessment data), All ages pooled.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - PXVX0317 | Group 2 - Placebo
Number analyzed (Participants) | 206 | 207
Participants | 0 | 1

8. Secondary Outcome: Anti-CHIKV SNA Titer (NT80) Seroresponse Rates at Days 15 and 183
Description: Difference in anti-CHIKV SNA titer (NT80) seroresponse rate (PXVX0317 minus placebo) with associated 95 percent CIs at Day 15 and Day 183.
Time Frame: Day 15 and 183 (14 and 182 days postvaccination, respectively)
Population: Immunogenicity evaluable population (all randomized and vaccinated participants who provided an evaluable Day 22 anti-CHIKV human SNA assay sample within the analysis window, had no measurable anti-CHIKV human SNA assay titer at Day 1, and had no important protocol deviation deemed exclusionary or other reason to be excluded as defined prior to unblinding).
  Number analyzed is number of participants with a sample result available at the indicated visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 - PXVX0317 | Group 2 - Placebo
Number analyzed (Participants) | 189 | 183
percentage of participants
  Day 15: number analyzed (Participants) | 181 | 176
  Day 15 | 82.3 [76.1 to 87.2] | 2.8 [1.2 to 6.5]
  Day 183: number analyzed (Participants) | 184 | 173
  Day 183 | 75.5 [68.9 to 81.2] | 1.2 [0.3 to 4.1]
Statistical Analysis 1: Comparison: Group 1 - PXVX0317 vs Group 2 - Placebo; Day 15; Test type: Superiority; p < 0.0001, Chi-squared — Key secondary endpoints were tested hierarchically (Day 15 tested prior to Day 183), such that each was only tested if both coprimary endpoints and prior key secondary endpoints were met, so no multiple comparisons were performed; p-value is from a two-sided chi-square test of equality of seroresponse percentages between groups; Percent Difference = 79.5, 95% CI 2-sided [72.3 to 84.6] — Seroresponse rate difference is (PXVX0317 minus placebo)
Statistical Analysis 2: Comparison: Group 1 - PXVX0317 vs Group 2 - Placebo; Day 183; Test type: Superiority; p < 0.0001, Chi-squared — [p-value comment as in outcome 8, analysis 1]; p-value is from a two-sided chi-square test of equality of seroresponse percentages between groups; Percent Difference = 74.4, 95% CI 2-sided [67.1 to 80.1] — Seroresponse rate difference is (PXVX0317 minus placebo)

9. Secondary Outcome: Anti-CHIKV SNA GMTs at Days 15 and 183
Description: Anti-CHIKV SNA GMTs with associated 95 percent CIs at Day 15, and Day 183 for PXVX0317 (CHIKV VLP vaccine) and placebo for the IEP, all age strata combined.
Time Frame: Day 15, and 183 (14 and 182 days postvaccination, respectively)
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1 - PXVX0317 | Group 2 - Placebo
Number analyzed (Participants) | 189 | 183
Titer
  Day 15: number analyzed (Participants) | 181 | 176
  Day 15 | 378 [301 to 476] | 9 [7 to 11]
  Day 183: number analyzed (Participants) | 184 | 173
  Day 183 | 233 [194 to 280] | 8 [7 to 10]
Statistical Analysis 1: Comparison: Group 1 - PXVX0317 vs Group 2 - Placebo; Day 15; Test type: Superiority; p < 0.0001, ANOVA; [statistical method as in outcome 2, analysis 1]; [GMT Ratio] = 42, 95% CI 2-sided [32 to 56] — Ratio of GMTs is (PXVX0317:placebo)
Statistical Analysis 2: Comparison: Group 1 - PXVX0317 vs Group 2 - Placebo; Day 183; Test type: Superiority; p < 0.0001, ANOVA; [statistical method as in outcome 2, analysis 1]; [GMT Ratio] = 28, 95% CI 2-sided [22 to 35] — Ratio of GMTs is (PXVX0317:placebo)

10. Secondary Outcome: Anti-CHIKV SNA Geometric Mean Fold Increase (GMFI)
Description: Geometric mean fold increase (GMFI) in anti-CHIKV SNA titers from Day 1 to Day 15, Day 22, and Day 183 for the IEP for all age strata combined.
Time Frame: Day 15, 22, and 183 (14, 21 and 182 days postvaccination, respectively)
Population: Immunogenicity evaluable population (all randomized and vaccinated participants who provided an evaluable Day 22 anti-CHIKV human SNA assay sample within the analysis window, had no measurable anti-CHIKV human SNA assay titer at Day 1, and had no important protocol deviation deemed exclusionary or other reason to be excluded as defined prior to unblinding).
  Number analyzed is number of participants with a sample result available at both Day 1 and the indicated visit.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase in Anti-CHIKV SNA titre
Arm/Group | Group 1 - PXVX0317 | Group 2 - Placebo
Number analyzed (Participants) | 189 | 183
Fold increase in Anti-CHIKV SNA titre
  Day 15: number analyzed (Participants) | 181 | 176
  Day 15 | 48.5 [40.1 to 58.7] | 1.2 [1.0 to 1.4]
  Day 22 | 93.9 [78.0 to 113.1] | 1.1 [0.9 to 1.3]
  Day 183: number analyzed (Participants) | 184 | 173
  Day 183 | 29.3 [25.0 to 34.4] | 1.0 [0.9 to 1.2]
Statistical Analysis 1: Comparison: Group 1 - PXVX0317 vs Group 2 - Placebo; Day 15; Test type: Superiority; p < 0.0001, t-test, 2 sided — GMFI estimates and 95 percent CIs are based on t-statistics assuming a normal distribution of the log fold increase in titer. p-value tests equality of log fold increase in titer between groups
Statistical Analysis 2: Comparison: Group 1 - PXVX0317 vs Group 2 - Placebo; Day 22; Test type: Superiority; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Group 1 - PXVX0317 vs Group 2 - Placebo; Day 183; Test type: Superiority; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 10, analysis 1]

11. Secondary Outcome: Subjects With Anti-CHIKV SNA Titer ≥15 and 4-fold Rise Over Baseline
Description: Number and percentage of participants with anti-CHIKV SNA titers ≥15 and 4-fold rise over baseline at Day 15, Day 22, and Day 183 for the IEP for all age strata combined.
Time Frame: Day 15, 22 and 183 (14, 21 and 182 days postvaccination, respectively)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 - PXVX0317 | Group 2 - Placebo
Number analyzed (Participants) | 189 | 183
percentage of participants
  SNA titers ≥ 15 at Day 15: number analyzed (Participants) | 181 | 176
  SNA titers ≥ 15 at Day 15 | 94.5 [90.1 to 97.0] | 2.8 [1.2 to 6.5]
  SNA titers ≥ 15 at Day 22 | 95.2 [91.2 to 97.5] | 1.1 [0.3 to 3.9]
  SNA titers ≥ 15 at Day 183: number analyzed (Participants) | 184 | 173
  SNA titers ≥ 15 at Day 183 | 92.9 [88.3 to 95.8] | 1.2 [0.3 to 4.1]
  ≥4-fold rise over baseline at Day 15: number analyzed (Participants) | 181 | 176
  ≥4-fold rise over baseline at Day 15 | 85.6 [79.8 to 90.0] | 2.8 [1.2 to 6.5]
  ≥4-fold rise over baseline at Day 22 | 89.4 [84.2 to 93.0] | 1.1 [0.3 to 3.9]
  ≥4-fold rise over baseline at Day 183: number analyzed (Participants) | 184 | 173
  ≥4-fold rise over baseline at Day 183 | 83.2 [77.1 to 87.9] | 1.2 [0.3 to 4.1]
Statistical Analysis 1: Comparison: Group 1 - PXVX0317 vs Group 2 - Placebo; SNA titers ≥15 at Day 15; Test type: Superiority; p < 0.0001, Chi-squared; p-value is from a two-sided chi-square test of equality of SNA response percentages between groups; Percent Difference = 91.6, 95% CI 2-sided [86.0 to 94.6] — SNA response rate difference is (PXVX0317 minus placebo)
Statistical Analysis 2: Comparison: Group 1 - PXVX0317 vs Group 2 - Placebo; SNA titers ≥15 at Day 22; Test type: Superiority; p < 0.0001, Chi-squared; p-value is from a two-sided chi-square test of equality of seroresponse percentages between groups; Percent Difference = 94.1, 95% CI 2-sided [89.2 to 96.5] — Seroresponse rate difference is (PXVX0317 minus placebo)
Statistical Analysis 3: Comparison: Group 1 - PXVX0317 vs Group 2 - Placebo; SNA titers ≥15 at Day 183; Test type: Superiority; p < 0.0001, Chi-squared; p-value is from a two-sided chi-square test of equality of SNA response percentages between groups; Percent Difference = 91.8, 95% CI 2-sided [86.3 to 94.8] — SNA response rate difference is (PXVX0317 minus placebo)
Statistical Analysis 4: Comparison: Group 1 - PXVX0317 vs Group 2 - Placebo; ≥4-fold rise over baseline at Day 15; Test type: Superiority; p < 0.0001, Chi-squared — p-value is from a two-sided chi-square test of equality of SNA response percentages between groups; Percent Difference = 82.8, 95% CI 2-sided [75.9 to 87.5] — SNA response rate difference is (PXVX0317 minus placebo)
Statistical Analysis 5: Comparison: Group 1 - PXVX0317 vs Group 2 - Placebo; ≥4-fold rise over baseline at Day 22; Test type: Superiority; p < 0.0001, Chi-squared; p-value is from a two-sided chi-square test of equality of SNA response percentages between groups; Percent Difference = 88.3, 95% CI 2-sided [82.4 to 92.0] — SNA response rate difference is (PXVX0317 minus placebo)
Statistical Analysis 6: Comparison: Group 1 - PXVX0317 vs Group 2 - Placebo; ≥4-fold rise over baseline at Day 183; Test type: Superiority; p < 0.0001, Chi-squared; p-value is from a two-sided chi-square test of equality of SNA response percentages between groups; Percent Difference = 82.0, 95% CI 2-sided [75.2 to 86.8] — SNA response rate difference is (PXVX0317 minus placebo)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Day 1 through to the Day 183 end of study visit.
Description: A solicited AE is a protocol-specified AE about which the investigator (or designee) proactively asks the participants during a protocol-specified time period. A reactogenicity event may be considered as a solicited AE per discretion of the investigator. (Systematic Assessment)
  An unsolicited AE is an AE that is spontaneously reported by the participant or discovered by the investigator (Non-systematic Assessment).
Arm/Group | Group 1 - PXVX0317 | Group 2 - Placebo
All-Cause Mortality (participants affected / at risk) | 1/206 | 1/207
Serious Adverse Events (participants affected / at risk) | 4/206 | 3/207
Other Adverse Events (participants affected / at risk) | 46/206 | 44/207
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - PXVX0317 (N=206) | Group 2 - Placebo (N=207)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - PXVX0317 (N=206) | Group 2 - Placebo (N=207)
Fatigue (General disorders) | 13 (13) | 12 (12)
Headache (Nervous system disorders) | 9 (9) | 16 (16)
Myalgia (Musculoskeletal and connective tissue disorders) | 13 (13) | 13 (13)
Injection Site Pain (General disorders) | 11 (11) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This is a multi-center study and agreement with investigators depends on the individual site contact.

DOCUMENTS (2):
  • Study Protocol (2023-03-31): https://cdn.clinicaltrials.gov/large-docs/17/NCT05349617/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-31): https://cdn.clinicaltrials.gov/large-docs/17/NCT05349617/SAP_001.pdf